CLINICAL TRIAL: NCT05372003
Title: IL-4 & Insulin Resistance in Patients With Atopic Dermatitis
Brief Title: IL-4 and Insulin Resistance for Treatment of Patients With Atopic Dermatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elena Anna (Eleanna) De Filippis, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-002567
Record Dates: First submitted 2022-04-29; First posted 2022-05-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects on Dupilumab (Experimental): individuals with atopic dermatitis placed on dupilumab for more than 6 months will be eligible to this study. Their metabolic profile will be compared to the group of "Subjects on Phototherapy"
  Interventions: Drug: Dupilumab
- Subjects on Phototherapy (Active Comparator): individuals with atopic dermatitis placed on phototherapy for more than 6 months will be eligible to this study to serve as an active comparator to the "Subjects with Dupilumab"
  Interventions: Other: Photo therapy

INTERVENTIONS:
Drug: Dupilumab — dupilumab injections will be prescribed and managed by dermatology as standard of care
  Arms: Subjects on Dupilumab
Other: Photo therapy — light therapy will be prescribed and managed by dermatology as standard of care
  Other Names: light therapy
  Arms: Subjects on Phototherapy

SUMMARY:
The purpose of this study is to better understand the interactions between the innate immune system, in particular eosinophils, their secreted cytokines (interleukin-4), and metabolism in human health and disease states such as obesity and insulin resistance.

DETAILED DESCRIPTION:
Patients with a body mass index (BMI) less than 30 kg/m2 and a history of atopic dermatitis on long-term (greater than 6 months) treatment with dupilumab. Researchers will compare in vivo evaluations of insulin sensitivity in subjects on dupilumab vs subjects matched for similar weight and BMI, with atopic dermatitis, but without dupilumab therapy (phototherapy).

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign informed consent form.
* Body mass index (BMI), 22-29 kg/m^2.
* Diagnosis of Atopic Dermatitis treated with dupilumab for longer than 6 months.
* Diagnosis of Atopic Dermatitis treated with topical steroids or phototherapy.

Exclusion Criteria:

* Any prescription for systemic glucocorticoid, immunosuppressant, antidiabetic medications in the past 6 months.
* Evidence of diabetes mellitus.
* Morning Cortisol < 5 mg/dl (collected before 10.30 am).
* Presence of acute illness.
* Low hemoglobin or hematocrit.
* Current participation in a weight-loss regimen, with a weight loss > 10% total body weight in the last 6 months).
* Smoking history in the last 6 months (tobacco, nicotine-containing products including e-cigarettes).
* Pregnant or breastfeeding.
* Personal history of gastric bypass surgery.
* Previous participation in a clinical trial with an investigational product in the past 30 days, or 5 half-lives, or twice the duration of the biological effect of the investigational drug (whichever is longest).
* Exposed to more than 4 new chemical entities within 12 months before study enrollment.
* Any other condition or event considered exclusionary by the PI and the study physician.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Homa IR | baseline
  Homeostatic Model Assessment of Insulin Resistance will be calculated by multiplying the fasting glucose concentration (mg/dl) by the fasting insulin concentration (mmol/L).
Matsuda Index | baseline
  The Matsuda index is able to estimate peripheral insulin sensitivity by computing the product of glucose and insulin collected during the OGTT.

SECONDARY OUTCOMES:
Adipo-IR | baseline
  Adipo-IR will be calculated by multiplying the fasting FFA concentration (mmol/L) by the fasting insulin concentration (pmol/L) obtained during the baseline blood collection during the oral glucose tolerance test
Systemic inflammatory markers | baseline
  Circulating plasma levels of inflammatory markers interleukin 1 (IL1), Tumor necrosis factor alpha (TNFa), highly sensitive C-reactive protein (hs-CRP), Monocyte Chemoattractant Protein 1 (MCP1), interleukin 6 (IL-6), Interleukin 4 (IL-4) and interleukin 13 (IL13)
Adipokines | baseline
  We will measure the plasma levels of adipokines (leptin and adiponectin) by radioimmunoassay and ELISA in all subjects recruited and compared across study group
Fasting Free Fatty Acid | baseline
  During the OGTT, we will collect fasting blood to assess levels of plasma free fatty acid (mmol/L). These values will be compared across the 2 different group studied.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Anna De Filippis, MD, PhD, Principal Investigator — Mayo
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials